CLINICAL TRIAL: NCT04144686
Title: 'Effectiveness of Customised Vestibular Rehabilitation With and Without Additional Dual-Task Training in Persons With a Chronic Vestibular Disorder. A Randomised Controlled Trial'
Brief Title: Advances in Vestibular Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19/LO/1066
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-07

CONDITIONS: Vestibular
Keywords: Vestibular; dual-tasking; Gait; rehabilitation; dizziness
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Intervention Model Description: Single Blinded Randomised Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: This RCT has a single mask (assessor blinded). The blinded outcome assessors will collect all the outcome measure data at baseline (week 0) and follow-up (week 6 and 12). The outcome assessor will be asked to record any incidences of unblinding and how this occurred. Blinded outcome assessors will all be trained by Dr Marousa Pavlou or Ms Viktoria Azoidou on how to complete all assessments for parity. During the course of the study, blinded assessors will be MSc students who will work on the project as part of their MSc thesis or other PhD students in the department.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Vestibular participants undertaking a single-task vestibular rehabilitation
  Interventions: Other: Physiotherapy Rehabilitation
- Group B (Experimental): Vestibular participants undertaking a dual-task vestibular rehabilitation
  Interventions: Other: Physiotherapy Rehabilitation

INTERVENTIONS:
Other: Physiotherapy Rehabilitation — Participants will be randomly allocated, using a random number generator, to a 12-week supervised customised exercise group incorporating VRT programme without (Group A) or with cognitive DT exercises (Group B).

SUMMARY:
Vestibular rehabilitation therapy (VRT) is an exercise-based programme to encourage central nervous system (CNS) compensation for vestibular dysfunction. There is moderate to strong evidence to support VRT as a safe, effective management in reducing dizziness, vertigo, associated falls and improving quality of life in people with a unilateral and bilateral peripheral vestibular disorder. However, the evidence to discriminate between differing forms of treatment is unclear and, although, approximately 50% to 80% of persons with a vestibular dysfunction achieve significant subjective symptom, gait, dynamic visual acuity and postural stability improvements, full recovery is less common for reasons that currently remain unknown. Thus, further studies are required to identify optimal VRT approaches.

The purpose of this investigation is to identify if the incorporation of dual-task (DT) exercises into a customised VRT programme will have an effect on treatment outcomes in persons with chronic vestibular disorders.

DETAILED DESCRIPTION:
The vestibular system system (i.e. inner ear balance system) is responsible for sending information to the brain about how fast our head is moving as well as about static head position, is necessary for us to be able to see clearly when turning our heads, to navigate in the dark and to balance. Persons who have an inner ear balance disorder will commonly report subjective symptoms of dizziness, imbalance, blurry vision, difficulty concentrating, imbalance and increased falls. Customised vestibular rehabilitation is the mainstay of treatment for persons with an inner ear balance disorder. Eye, head and body movement exercises are included (i.e. walking while turning your head left and right to scan the road) as appropriate for each individual. Moderate to strong evidence exists to support vestibular rehabilitation as a safe, effective management for persons with an inner ear balance disorder. However, there is insufficient evidence to discriminate between differing forms of treatment and although approximately 50% to 80% of persons with a vestibular dysfunction achieve significant symptomatic (i.e. dizziness) and objective improvements with regards to their balance, walking and activities of daily living, some persons do not improve. The reasons for this remain unclear. Thus, although vestibular rehabilitation has been shown to be safe and effective, further studies are required to identify optimal vestibular rehabilitation treatment approaches. Dual-task training (i.e. simultaneously performing two different activities such as walking and talking) has been shown to be beneficial in improving balance and complex walking ability (i.e. walking with head turns) in older adults. However, no studies have investigated dual-tasking training in persons with a vestibular disorder. This is despite evidence showing that the ability to perform complex walking tasks is negatively affected in persons with a vestibular disorder when a cognitive (i.e. "thinking") task is added. Therefore, the purpose of this study is to compare the effect of customised vestibular rehabilitation with and without the incorporation of dual-task (DT) exercises on subjective symptom, objective complex walking tasks, "thinking" function and psychological state. The hypothesis is that customised vestibular rehabilitation incorporating DT exercises will provide greater benefit compared to customised vestibular rehabilitation in isolation.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of a peripheral vestibular disorder
* chronic dizziness and/or unsteadiness
* 18 to 80 years' old
* previous vestibular rehabilitation programme completed with partial/no improvement
* willing to participate and to comply with the proposed training and testing regime

Exclusion Criteria:

Persons with

* central nervous system involvement, excluding migraine
* fluctuating symptoms, for example, active Ménière disease
* acute orthopaedic disorders influencing balance control and gait
* a score of < 23/30 on the MoCA
* a score of >15/21 on the HADS for the depression component indicating significant depression symptoms
* inability to attend sessions
* lack of a good grasp of written/spoken English will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Functional Gait Assessment | 10 minutes
  The primary outcome is the Functional Gait Assessment which is a 10-item test that assesses performance on complex gait tasks (i.e. walking with head turns, stepping over an obstacle or stopping and turning). Scores range from 0 to 30. The highest score is 30 and greater outcomes are indicative of better performance while lower scores are indicative of poorer performance. The Functional Gait Assessment has been validated in healthy people, older adults with a history of falls and balance impairments, and people with a vestibular disorder. The minimal detectable change for Functional Gait Assessment is reported to be 6 points in persons with balance and vestibular disorders. Scores ≤22/30 identify fall risk and are predictable of falls in community-living older persons within 6 months.

SECONDARY OUTCOMES:
Functional Gait Dual-Task Test | 45 minutes
  The FGA in isolation will always be completed first in (primary outcome measure), followed by the dual-task (DT) test conditions, which will be completed in random order. The cognitive DT condition will involve a numeracy and literacy task and the auditory stimuli will involve restaurant noise.
Mini-Balance Evaluation Systems Test | 10 minutes
  The Mini-Balance Evaluation Test is a measure of dynamic balance (anticipatory postural adjustments, reactive postural control, sensory orientation and dynamic gait). The Mini-Balance Evaluation Systems Test consists of 14 items, with scores ranging from 0 to 28 points. Higher scores indicate better outcome while lower scores poorer outcome. Scores ≤ 20/32 indicate increased falls risk.
Cambridge Neuropsychological Test Automated Battery | 50 minutes
  Cambridge Neuropsychological Test Automated Battery is a semiautomated computer program that utilizes a touch screen technology and press pad, to assess neurocognitive function. The Cambridge Neuropsychological Test Automated Battery core cognition battery is a validated cognitive assessment system for assessing multiple components of cognitive function, including attention, visual memory, spatial memory, executive function and reaction time.
Montreal Cognitive Assessment Tool | 5 minutes
  The Montreal Cognitive Assessment Tool is a rapid screening tool for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive function, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The scores range from 0-30. Higher scores indicate better outcomes while lower scores are indicative of poorer outcomes. It has been recommended that a cut-off scores of 23/30 be used to identify multi-domain cognitive impairment.
Speech in Babble Test | 10 minutes
  The Speech in Babble Test is a low redundancy speech in babble type noise test. The Speech in Babble Test is presented on a calibrated computer using Matlab software. There are 8 in total phonemically and phonetically balanced word lists. The words are presented in the background of a 20-talker babble noise. Two randomly selected monosyllabic consonant vowel consonant word lists in a background of multitalker babble are presented to each ear (i.e. each ear is tested twice). The signal to noise ratio during the test is varied adaptively.
Standard pure tone audiometry | 10 minutes
  Standard pure tone audiometry is considered a 'gold' standard test of audiologic examination. This test will be completed with a portable calibrated audiometer (GSI Pello Standard model with DD45's, IP30 and B81, Serial Number: GS0071085, calibrated by Guymark UK Ltd).
Axivity Wrist Band 3-Axis logging accelerometer | 7 days
  Participants' physical activity level will be assessed using a wrist-worn accelerometer, the Axivity Wrist Band 3-Axis logging accelerometer. The Axivity Wrist Band 3-Axis logging accelerometer captures triaxial acceleration data at 100 Hz with a dynamic range of ±8 g and has been widely used in population-based studies to assess physical activity levels.
Activity-specific Balance Confidence Scale | 3 minutes
  The Activity-specific Balance Confidence Scale is a self-perceived questionnaire with 16 items and assesses balance confidence in daily activities. Scores range from 0 to 100. Higher scores are indicative of better outcome while lower scores indicate poorer outcome. A score ≤67/100 indicate increased falls risk.
Hospital Anxiety and Depression Scale | 3 minutes
  The Hospital Anxiety and Depression Scale, a 14-item scale which assesses non-somatic anxiety and depression symptoms, will also be completed. Scores range from 0 to 21 for each subscale with a score ≥8 proposed for the identification of caseness, for both depression and anxiety. Higher scores are indicative of poorer outcomes.
Pittsburgh Sleep Quality Index | 3 minutes
  The Pittsburgh Sleep Quality Index generates seven component scores: subjective sleep quality, sleep latency, sleep duration habitual sleep efficiency, sleep disturbance, use of sleeping medication, and daytime dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality while lower scores indicate better outcomes. In distinguishing good and poor sleepers, a global Pittsburgh Sleep Quality Index score >5 yields a sensitivity of 89.6% and a specificity of 86.5%.
Epworth Sleepiness Scale | 3 minutes
  The Epworth Sleepiness Scale is a validated and widely used questionnaire exploring daytime sleepiness. It consists of eight questions that are added together to obtain a single number. Higher scores indicate sleeping disorder while lower scores are indicative of better outcomes. Scores range from 0 to 24. The reference range of 'normal' Epworth Sleepiness Scale scores is 0-10 while Epworth Sleepiness Scale scores of 11-24 represent increasing levels of 'excessive daytime sleepiness'.
EQ-5D-5L | 3 minutes
  The EQ-5D-5L is a generic measure of health status for clinical and economic appraisal. The EQ-5D-5L descriptive system comprises of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.
Vertigo Symptom Scale | 3 minutes
  The VSS is used to assess the frequency and severity of common vestibular (Vertigo Symptom Scale-V; e.g. vertigo, imbalance) and autonomic/somatic (Vertigo Symptom Scale-A; e.g. heart pounding, heavy feeling in the arms or legs) symptoms. Scores range from 0 to 60. Normalised scores range from 0-4, with higher scores indicating a higher (i.e. worse) level of symptoms while lower scores indicate better outcomes.
Situational Vertigo Questionnaire | 3 minutes
  The Situational Vertigo Questionnaire -shortened version measures how frequently symptoms are provoked or exacerbated in environments with visual vestibular mismatch or intense visual motion (e.g. travelling on escalators, crowds, scrolling computer screens). Scores range from 0 to 4. Higher scores indicate poorer outcomes while lower scores are indicative of better outcomes. Scores ≥0.7/4 indicate visual induced dizziness symptoms.
Dizziness Handicap Inventory | 3 minutes
  The Dizziness Handicap Inventory is a 25-item self-assessment inventory designed to evaluate self-perceived handicap imposed by symptoms of dizziness. It consists of three domains: emotional, functional and physical. Total scores range from 0 to 100, with higher score indicating greater perceived handicap while lower scores are indicative of better performance. Scores between 0-30, 31-60, and 61-100 on the Dizziness Handicap Inventory indicate mild, moderate, and severe perceived handicap respectively, and can differentiate a person's functional abilities.
Cognitive and Behavioural Symptom Questionnaire | 3 minutes
  The Cognitive and Behavioural Symptom Questionnaire is a measure of subjects' cognitive (i.e. beliefs) and behavioural responses to symptoms of their health condition. This measure includes five cognitive (i.e. beliefs) subscales: Symptom Focusing, Catastrophizing, Damaging Beliefs, Fear Avoidance and Embarrassment Avoidance; and two behavioural subscales: All or- Nothing and Avoidance/Rest.
The Illness Perception Questionnaire-Revised | 3 minutes
  The Illness Perception Questionnaire-Revised was used to measure participants' illness perceptions. The Illness Perception Questionnaire-Revised measures the key components in Leventhal's common sense self-regulatory model: Illness identity will measured by asking patients to indicate whether they have experienced and attribute a number of potential symptoms to their dizziness condition. Scores range from 0 to 24 with higher scores indicating increased illness identity while lower scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Viktoria Azoidou, Principal Investigator — Ms
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will be processed in accordance with the General Data Protection Regulation 2016 (GDPR). All information collected will be kept strictly confidential and stored anonymously on password protected computers used only by research staff. Data will be stored securely in accordance with the Data Protection Act (1998) and the General Data Protection Regulations which came into effect on 25 May 2018. IPD will not be passed on to anyone outside of participant's medical care team. Stored, anonymised data may be used for future medical and health-related studies. IPD will be retained for 10 years after it has been collected.

REFERENCES:
- [Result] Hall CD, Herdman SJ, Whitney SL, Cass SP, Clendaniel RA, Fife TD, Furman JM, Getchius TS, Goebel JA, Shepard NT, Woodhouse SN. Vestibular Rehabilitation for Peripheral Vestibular Hypofunction: An Evidence-Based Clinical Practice Guideline: FROM THE AMERICAN PHYSICAL THERAPY ASSOCIATION NEUROLOGY SECTION. J Neurol Phys Ther. 2016 Apr;40(2):124-55. doi: 10.1097/NPT.0000000000000120. PMID 26913496
- [Result] Smith PF. Age-Related Neurochemical Changes in the Vestibular Nuclei. Front Neurol. 2016 Mar 3;7:20. doi: 10.3389/fneur.2016.00020. eCollection 2016. PMID 26973593
- [Result] Topuz O, Topuz B, Ardic FN, Sarhus M, Ogmen G, Ardic F. Efficacy of vestibular rehabilitation on chronic unilateral vestibular dysfunction. Clin Rehabil. 2004 Feb;18(1):76-83. doi: 10.1191/0269215504cr704oa. PMID 14763722
- [Result] Arnold SA, Stewart AM, Moor HM, Karl RC, Reneker JC. The Effectiveness of Vestibular Rehabilitation Interventions in Treating Unilateral Peripheral Vestibular Disorders: A Systematic Review. Physiother Res Int. 2017 Jul;22(3). doi: 10.1002/pri.1635. Epub 2015 Jun 25. PMID 26111348
- [Result] Lacour M, Bernard-Demanze L, Dumitrescu M. Posture control, aging, and attention resources: models and posture-analysis methods. Neurophysiol Clin. 2008 Dec;38(6):411-21. doi: 10.1016/j.neucli.2008.09.005. Epub 2008 Oct 9. PMID 19026961
- [Result] Yogev-Seligmann G, Hausdorff JM, Giladi N. The role of executive function and attention in gait. Mov Disord. 2008 Feb 15;23(3):329-42; quiz 472. doi: 10.1002/mds.21720. PMID 18058946
- [Result] Carson N, Leach L, Murphy KJ. A re-examination of Montreal Cognitive Assessment (MoCA) cutoff scores. Int J Geriatr Psychiatry. 2018 Feb;33(2):379-388. doi: 10.1002/gps.4756. Epub 2017 Jul 21. PMID 28731508
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Result] Davies RA, Luxon LM. Dizziness following head injury: a neuro-otological study. J Neurol. 1995 Mar;242(4):222-30. doi: 10.1007/BF00919595. PMID 7798121
- [Result] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Result] Lempert T, Olesen J, Furman J, Waterston J, Seemungal B, Carey J, Bisdorff A, Versino M, Evers S, Newman-Toker D. Vestibular migraine: diagnostic criteria. J Vestib Res. 2012;22(4):167-72. doi: 10.3233/VES-2012-0453. PMID 23142830
- [Result] Neuhauser H, Leopold M, von Brevern M, Arnold G, Lempert T. The interrelations of migraine, vertigo, and migrainous vertigo. Neurology. 2001 Feb 27;56(4):436-41. doi: 10.1212/wnl.56.4.436. PMID 11222783
- [Result] Wrisley DM, Marchetti GF, Kuharsky DK, Whitney SL. Reliability, internal consistency, and validity of data obtained with the functional gait assessment. Phys Ther. 2004 Oct;84(10):906-18. PMID 15449976
- [Result] Marchetti GF, Lin CC, Alghadir A, Whitney SL. Responsiveness and minimal detectable change of the dynamic gait index and functional gait index in persons with balance and vestibular disorders. J Neurol Phys Ther. 2014 Apr;38(2):119-24. doi: 10.1097/NPT.0000000000000015. PMID 24637931
- [Result] Wrisley DM, Kumar NA. Functional gait assessment: concurrent, discriminative, and predictive validity in community-dwelling older adults. Phys Ther. 2010 May;90(5):761-73. doi: 10.2522/ptj.20090069. Epub 2010 Apr 1. PMID 20360052
- [Result] Godi M, Franchignoni F, Caligari M, Giordano A, Turcato AM, Nardone A. Comparison of reliability, validity, and responsiveness of the mini-BESTest and Berg Balance Scale in patients with balance disorders. Phys Ther. 2013 Feb;93(2):158-67. doi: 10.2522/ptj.20120171. Epub 2012 Sep 27. PMID 23023812
- [Result] Leddy AL, Crowner BE, Earhart GM. Utility of the Mini-BESTest, BESTest, and BESTest sections for balance assessments in individuals with Parkinson disease. J Neurol Phys Ther. 2011 Jun;35(2):90-7. doi: 10.1097/NPT.0b013e31821a620c. PMID 21934364
- [Result] King L, Horak F. On the mini-BESTest: scoring and the reporting of total scores. Phys Ther. 2013 Apr;93(4):571-5. doi: 10.2522/ptj.2013.93.4.571. No abstract available. PMID 23547173
- [Result] Cambridge-Cognition-Limited. CANTABeclipse™: Test Administration Guide Manual. 3rd ed. Cambridge 2015.
- [Result] Egerhazi A, Berecz R, Bartok E, Degrell I. Automated Neuropsychological Test Battery (CANTAB) in mild cognitive impairment and in Alzheimer's disease. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Apr 13;31(3):746-51. doi: 10.1016/j.pnpbp.2007.01.011. Epub 2007 Jan 16. PMID 17289240
- [Result] Fowler KS, Saling MM, Conway EL, Semple JM, Louis WJ. Paired associate performance in the early detection of DAT. J Int Neuropsychol Soc. 2002 Jan;8(1):58-71. PMID 11843075
- [Result] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Result] Bamiou DE, Iliadou VV, Zanchetta S, Spyridakou C. What Can We Learn about Auditory Processing from Adult Hearing Questionnaires? J Am Acad Audiol. 2015 Nov-Dec;26(10):824-37. doi: 10.3766/jaaa.15009. PMID 26554488
- [Result] British Society of Audiology. Standard pure tone audiometry. British Society of Audiology-BSA 2017.
- [Result] British Society of Audiology. Standard pure tone audiometry. British Society of Audiology-BSA 2011.
- [Result] Doherty A, Jackson D, Hammerla N, Plotz T, Olivier P, Granat MH, White T, van Hees VT, Trenell MI, Owen CG, Preece SJ, Gillions R, Sheard S, Peakman T, Brage S, Wareham NJ. Large Scale Population Assessment of Physical Activity Using Wrist Worn Accelerometers: The UK Biobank Study. PLoS One. 2017 Feb 1;12(2):e0169649. doi: 10.1371/journal.pone.0169649. eCollection 2017. PMID 28146576
- [Result] Lee IM, Shiroma EJ. Using accelerometers to measure physical activity in large-scale epidemiological studies: issues and challenges. Br J Sports Med. 2014 Feb;48(3):197-201. doi: 10.1136/bjsports-2013-093154. Epub 2013 Dec 2. PMID 24297837
- [Result] Clarke CL, Taylor J, Crighton LJ, Goodbrand JA, McMurdo MET, Witham MD. Validation of the AX3 triaxial accelerometer in older functionally impaired people. Aging Clin Exp Res. 2017 Jun;29(3):451-457. doi: 10.1007/s40520-016-0604-8. Epub 2016 Jul 19. PMID 27435918
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Result] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Result] Yardley L, Masson E, Verschuur C, Haacke N, Luxon L. Symptoms, anxiety and handicap in dizzy patients: development of the vertigo symptom scale. J Psychosom Res. 1992 Dec;36(8):731-41. doi: 10.1016/0022-3999(92)90131-k. PMID 1432863
- [Result] Guerraz M, Yardley L, Bertholon P, Pollak L, Rudge P, Gresty MA, Bronstein AM. Visual vertigo: symptom assessment, spatial orientation and postural control. Brain. 2001 Aug;124(Pt 8):1646-56. doi: 10.1093/brain/124.8.1646. PMID 11459755
- [Result] Bisdorff A, Von Brevern M, Lempert T, Newman-Toker DE. Classification of vestibular symptoms: towards an international classification of vestibular disorders. J Vestib Res. 2009;19(1-2):1-13. doi: 10.3233/VES-2009-0343. No abstract available. PMID 19893191
- [Result] Jacobson GP, Newman CW. The development of the Dizziness Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1990 Apr;116(4):424-7. doi: 10.1001/archotol.1990.01870040046011. PMID 2317323
- [Result] Whitney SL, Wrisley DM, Brown KE, Furman JM. Is perception of handicap related to functional performance in persons with vestibular dysfunction? Otol Neurotol. 2004 Mar;25(2):139-43. doi: 10.1097/00129492-200403000-00010. PMID 15021773
- [Result] Skerrett TN, Moss-Morris R. Fatigue and social impairment in multiple sclerosis: the role of patients' cognitive and behavioral responses to their symptoms. J Psychosom Res. 2006 Nov;61(5):587-93. doi: 10.1016/j.jpsychores.2006.04.018. PMID 17084135
- [Result] Moss-Morris R, Weinman J, Petrie KJ et al. The Revised Illness Perception Questionnaire (IPR-Q). Psychol Health 2002; 17(1): 1-16.
- [Result] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Result] Lajoie Y, Gallagher SP. Predicting falls within the elderly community: comparison of postural sway, reaction time, the Berg balance scale and the Activities-specific Balance Confidence (ABC) scale for comparing fallers and non-fallers. Arch Gerontol Geriatr. 2004 Jan-Feb;38(1):11-26. doi: 10.1016/s0167-4943(03)00082-7. PMID 14599700